CLINICAL TRIAL: NCT07006441
Title: The Effects of Preoperative and Postoperative Cardiac Rehabilitation in Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Cardiac Rehabilitation in Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Principal Investigator, Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: auhucgun04
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Bypass Graft Surgery; Coronary Artery Disease
Keywords: Coronary Artery Disease; Coronary Artery Bypass Graft Surgery; Preoperative Cardiac Rehabilitation; Postoperative Cardiac Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Preoperative cardiac rehabilitation + postoperative cardiac rehabilitation (structured exercise, respiratory physiotherapy, and patient education)
  Interventions: Other: Preoperative Cardiac Rehabilitation; Other: Postoperative Cardiac Rehabilitation
- Control Group (Active Comparator): Postoperative cardiac rehabilitation (structured exercise, respiratory physiotherapy, and patient education)
  Interventions: Other: Postoperative Cardiac Rehabilitation

INTERVENTIONS:
Other: Preoperative Cardiac Rehabilitation — Structured exercise program, respiratory physiotherapy, and patient education
  Arms: Experimental Group
Other: Postoperative Cardiac Rehabilitation — Structured exercise program, respiratory physiotherapy, and patient education

SUMMARY:
This randomized controlled trial investigates the comparative effects of a combined preoperative and postoperative cardiac rehabilitation program versus a postoperative-only program on functional capacity, pulmonary function, peripheral muscle strength, pain, kinesiophobia, and quality of life in patients undergoing coronary artery bypass graft (CABG) surgery. The study aims to determine whether initiating rehabilitation prior to surgery improves short-term postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone coronary artery bypass graft surgery
* Ejection Fraction (EF) > 40%
* Being between the ages of 18-65
* Being able to speak, read and understand in their own language
* Volunteering to participate in the study

Exclusion Criteria:

* Having an active or suspected infection
* Presence of an active tumour
* History of thrombophlebitis or pulmonary embolism within the last 3 months
* Having an orthopaedic, neurological or cardiovascular disease that may affect the assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | 2 weeks
  Forced Vital Capacity will be measured before six-minute walk test according to the guideline of ERS.
Forced Expiratory Volume in 1 second (FEV1) | 2 weeks
  Forced Expiratory Volume in 1 second will be measured before six-minute walk test according to the guideline of ERS.
Peak Expiratory Flow (PEF) | 2 weeks
  Peak Expiratory Flow will be measured before six-minute walk test according to the guideline of ERS.
Forced Expiratory Flow 25-75% (FEF25-75) | 2 weeks
  Forced Expiratory Flow 25-75% will be measured before six-minute walk test according to the guideline of ERS.
6-minute Walk Test | 2 weeks
  The 6-minute Walk Test will be performed according to ATS guidelines. Walking distance, minute ventilation, respiratory rate, inspiratory capacity and breathing reserve will be recorded.
M. Quadriceps Muscle Strength | 2 weeks
  The m. quadriceps muscle strength will be measured using the MicroFet 2 hand-held dynamometer (Hogan Health Industries, USA). The test will be repeated three times for the dominant side and the average value in kilograms (kg) will be recorded.
M. Biceps Muscle Strength | 2 weeks
  The m. biceps muscle strength will be measured using the MicroFet 2 hand-held dynamometer (Hogan Health Industries, USA). The test will be repeated three times for the dominant side and the average value in kilograms (kg) will be recorded.
Cough Peak Flow | 2 weeks
  Cough Peak Flow (CPF) will be measured using a peak expiratory flow meter. Participants will be instructed to take a maximal deep breath and then cough as forcefully as possible into the device; the highest value from three trials will be recorded in liters per minute (L/min). Measurements will be performed in a seated position, ensuring a tight mouth seal and consistent technique.

SECONDARY OUTCOMES:
Level of Pain | 2 weeks
  Pain assessment will be performed using the Visual Analog Scale (VAS) to evaluate chest pain levels. Participants will be asked to mark their current pain intensity on a 10 cm horizontal line, with "no pain" at one end and "worst imaginable pain" at the other. The distance in centimeters from the "no pain" end to the mark will be measured and recorded as the pain score.
Level of Fear of Movement | 2 weeks
  Fear of movement (kinesiophobia) will be assessed using the Tampa Scale for Kinesiophobia (TSK). Participants will complete the 17-item questionnaire, which evaluates fear of movement and re-injury on a 4-point Likert scale. The total score, ranging from 17 to 68, will be calculated, with higher scores indicating greater fear of movement.
Level of Quality of Life | 2 weeks
  Quality of life will be assessed using the Short Form-36 (SF-36) Health Survey. Participants will complete the 36-item questionnaire, which evaluates eight domains including physical functioning, bodily pain, general health, and mental well-being. Each domain will be scored from 0 to 100, with higher scores indicating better perceived quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Hikmet Ucgun, PT, PhD, Principal Investigator — Atlas University
Locations (1):
- Istanbul Atlas University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No